CLINICAL TRIAL: NCT04780165
Title: Prospective, Open Label, Multicenter Trial to Investigate the Efficacy and Tolerability of Blephademodex Wipes in Patients With Demodex Blepharitis
Brief Title: Efficacy and Tolerability of Blephademodex Wipes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LTPIVBDX19
Record Dates: First submitted 2020-09-23; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Demodex Blepharitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental)
  Interventions: Device: Blephademodex

INTERVENTIONS:
Device: Blephademodex — During the first 28 days of the trial, subjects will use one Blephademodex® eyelid hygiene wipe every evening per eye to clean the eyelids of both their eyes. At the start of the second period the Investigator will assess based on the GDS if the condition is resolved and manage accordingly: subjects will either continue with this regime if GDS is unchanged (further treatment phase) or revert to Blephaclean wipes every evening instead (maintenance phase), again to clean the eyelids of both their eyes.
  Other Names: Blephaclean

SUMMARY:
Primary Objective

- To evaluate efficacy of Blephademodex eyelid hygiene wipe treatment with a subsequent maintenance period with Blephaclean lid cleansing wipes in Demodex blepharitis, as assessed by the change in ocular symptoms by a Global Discomfort Scale (GDS).

Secondary Objectives

* To evaluate the efficacy of Blephademodex eyelid hygiene wipe treatment in Demodex blepharitis as assessed by the change alone and in combination with a subsequent maintenance period of treatment with Blephaclean eyelid cleansing wipes ocular symptoms by: adapted TOSS; SANDE; specific blepharitis symptoms; Demodex count; ocular surface redness (Efron scale); lid margin redness/swelling (Efron / custom scale); Dandruff coverage at bases of eyelashes; ocular surface staining (Oxford scale; corneal only)
* To evaluate subject and physician satisfaction with Blephademodex eyelid hygiene wipes
* To evaluate ease of use for Blephademodex eyelid hygiene wipes
* Adverse events are documented and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old, all genders
* Able to read, to write and to fully understand German language
* Good general health as determined by the investigator by medical history and physical appearance
* Provision of written informed consent prior to inclusion
* Moderate to Severe Blepharitis - grade ≥ 2 (Efron Scale)
* Global discomfort score (GDS) ≥ 4
* Proof of demodex infestation by at least ONE of the following:Demodex visible after lash manipulation;Cylindrical dandruff along the lash line; Lid margin itching; Madarosis

Exclusion Criteria:

* History of ocular trauma, ocular infection or intra-ocular inflammation within the 3 months before screening visit
* History of ocular refractive surgery and any other ocular surgeries within 3 months before screening visit
* History of ocular allergy or ocular herpes within the 3 months before screening visit
* History of inflammatory corneal ulcer within the 6 months before screening visit
* Sjogren syndrome or any other rheumatologic disease related dry eye
* Concurrent treatment with other eye drops (anti-infectives, steroids, prostaglandins (but artificial tears are ok).
* Specific Exclusion Criteria for Women:Patient who verbally confirms pregnancy or lactation; Childbearing potential woman who is not using a reliable method of contraception (oral contraceptive, intra-uterine device, subcutaneous contraceptive implant, vaginal ring, patch or condom) and is not surgically sterilised

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
Global Discomfort Score | Day 28
  Change from Baseline at Day 28 The Global (overall) discomfort score (GDS) consists of a single question, which can be answered by the subject by choosing a value between 0 (no discomfort) and 10 (worst discomfort): Thinking about today, how would you rate the discomfort of your eyes?
Global Discomfort Score | Day 56
  Change from D28 at Day 56

SECONDARY OUTCOMES:
Specific Blepharitis symptoms | Day 56
  Symptoms will be rated by the patient on the day of visit using 10-grade scales (0 = none to 10 = severe) for each of the following items Severity of any eyelid itching today / Severity of lid redness today / Severity of eyelid swelling today / How severe was the eyelid crusting this morning when you woke up? / How severe is missing lashes today?
adapted Total Ocular Symptom Score (TOSS) | Day 56
  8-item questionnaire with an overall score ranging from 0 ("none of the time") to 4 ("all of the time"). It contains of a single question concerning the frequency with which 8 different symptoms (itchy eyelids, eyelid redness, red eyes generally, swollen (puffy) eyes, tearing (eyes watering), crusting around the lashes, burning or stinging sensations and noticed eyelash loss) were experienced in the course of a week.
Symptom Assessment in Dry Eye (SANDE) | Day 56
  Comprised of two questions: 1) How often do your eyes feel dry and/or irritated? And 2) How severe you feel your symptoms of dryness and/or irritation are? This questionnaire uses a 100 mm horizontal line as visual analogue scale (VAS) for each question to assess ocular discomfort and/or dryness experienced by the patients. In the SANDE questionnaire, frequency of symptoms ranges from "rarely" to "all of the time" and the severity of symptoms ranges from "very mild" to "very severe".
Demodex count | Day 56
  Sideways 'pull' on 10 eyelashes - upper or lower lashes Extent (mites present? yes or no) and Severity/Intensity (1=1 tail; 2=2 tails; 3 =2+tails)
Ocular surface redness | Day 56
  Efron scale
Lid margin redness/swelling | Day 56
  Efron/custom scale
Cylindrical dandruff | Day 56
  Lash line coverage (%) and severity (mild/moderate/severe)
Ocular surface staining | Day 56
  Oxford scale; corneal only
Physician's impression and patient impression | Day 56
  Answer the item 'the treatment has been sufficiently effective' on a 4-point scale (strongly disagree, disagree, agree, strongly agree)
Tolerability of the wipes | Day 56
  Tolerability assessment by the physician and patient (0 = intolerable; 1 = somewhat tolerable; 2 = tolerable; 3 = fully tolerable)
Visual acuity | Day 56
  Snellen eye chart
Assessment of ease of use | Day 56
  as experienced by the subjects, rated on a five-point scale of "Very Difficult" to "Very Easy".

CONTACTS AND LOCATIONS:
Locations (1):
- Consultation office, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No